CLINICAL TRIAL: NCT03803787
Title: Prophylactic Inhaled Steroids to Reduce Radiation Pneumonitis Frequency and Severity in Non-small Cell Lung Cancer Patients
Brief Title: Prophylactic Inhaled Steroids to Reduce Radiation Pneumonitis Frequency and Severity in Lung Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Collaborators: Instituto Nacional de Enfermedades Respiratorias (Other Government)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, Head of the Thoracic Oncology unit, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CI/910/17
Record Dates: First submitted 2019-01-03; First posted 2019-01-15 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Radiation Pneumonitis
Keywords: Non-Small Cell Lung Cancer; Radiation Pneumonia; Lung cancer treatment; Respiratory Tract Neoplasms; Radiation fibrosis; Thoracic Neoplasms; Lung Diseases; Radiation Injury with Fibrosis; Radiation Fibrosis of Lung; Lung Injury
MeSH Terms: conditions — Radiation Pneumonitis; Carcinoma, Non-Small-Cell Lung; Respiratory Tract Neoplasms; Radiation Fibrosis Syndrome; Thoracic Neoplasms; Lung Diseases; Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- QT/RT + Budesonide (Experimental): Patients are receiving chemotherapy (QT) and radiotherapy (RT) plus inhaled Budesonide with space chamber at 400 mcg given twice daily initiating after the first dose of RT and continuing until pneumonitis development or 12 months completed.
  Interventions: Drug: Inhaled budesonide
- QT/RT + No medication (No Intervention): Patients are receiving chemotherapy (QT) and radiotherapy (RT) without intervention therapy and followed during 12 months.
- Target drug/RT + Budesonide (Experimental): Patients are receiving target therapy and radiotherapy (RT) plus inhaled Budesonide with space chamber at 400 mcg given twice daily initiating after the first dose of RT and continuing until pneumonitis development or 12 months completed.
  Interventions: Drug: Inhaled budesonide
- Target drug/RT + No medication (No Intervention): Patients are receiving target treatment and radiotherapy (RT) without intervention therapy and followed during 12 months.

INTERVENTIONS:
Drug: Inhaled budesonide — Patients will use inhaled budesonide (Numark) with space chamber at 400 mcg given twice daily initiating after the first dose of RT and continuing until pneumonitis development or 12 months completed.
  Other Names: Numark
  Arms: QT/RT + Budesonide; Target drug/RT + Budesonide

SUMMARY:
This randomized clinical study aims to assess whether prophylactic treatment with inhaled steroids in patients with locally advanced or concomitantly treated non-small cell lung carcinoma who are candidates for combination treatment with QT/RT or IMT + QT/RT.

The main questions it aims to answer are:

Whether prophylactic treatment decreases the severity of NPR on CTCAE v4.0 and RTOG scales.

Whether inhaled steroid use modifies the response to radiation therapy treatment compared to patients who do not receive prophylactic inhaled steroids.

DETAILED DESCRIPTION:
Clinical evaluation

The following BASELINE data shall be taken prior to radiation therapy:

Demographic, clinical, laboratory, and imaging data will be obtained from medical history and electronic records.

The patient will be instructed to perform the PFRs and tests of lung function.

Two EORTC, QLQ-C30, and QLQ LC13 quality of life questionnaires and three respiratory symptom questionnaires (St. George, dyspnea scale, and modified BORG) will be performed on the same day of lung function tests.

Additionally; blood samples will be taken for the evaluation of inflammatory mediators at the following times: BASAL (before RT), and every six weeks up to 48 weeks post-RT.

INTERVENTION GROUP

1. Prior to the onset of RT, the patient will be sorted to receive the control rather than experimental intervention (QT/RT or IMT + QT/RT) and a logbook to record adherence to treatment.
2. An IDM device shall be granted per month, containing the number of doses corresponding to 30 days. The record in the database of the day of the first session of RT will be taken to quantify the number of days of use of the drug and grant the next device per 30 days until the end of the study.
3. The patient will be instructed on the use of the device inhaled with the spacer chamber in the clinic Pulmonology consultation, alarm data and indications of the use of the drug will be given in writing, and knowledge will be reinforced at each visit.
4. The patient will be granted the drug use log where the patient will place the date and time of use of the drug to assess adherence to treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-small cell lung cancer (NSCLC) with unresectable locally advanced or metastatic disease (IIIA, IIIB or IV) of the classification tumor node, metastasis (TNM) of malignant lung tumors, 7th edition.
* NSCLC patients candidates for concomitant treatment (chemotherapy plus radiotherapy or target therapy plus radiotherapy).
* Evidence of measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2, Karnofsky 70-100.
* Life expectancy of > 4 months at the time of screening
* Patients with the ability to comply with the study and follow-up procedures.
* Patients with previous surgery less than four weeks.
* Must be willing and able to give signed informed consent and, in the opinion of the Investigator, to comply with the protocol tests and procedures.

Exclusion Criteria:

* Unstable systemic disease: active infection, heart, liver, kidney or metabolic disease; including uncontrolled chronic lung disease.
* Patients treated with systemic or inhaled corticosteroids.
* Patients of reproductive age without a family planning method, pregnant or lactating.
* Previous diagnosis of Pneumonitis with toxicity grade ≥ 2 by CTCAE v4.0 or RTOG scale.
* Patients with disease progression.
* Inspiratory flow < 90 liters / min.
* Discontinue of Treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pneumonitis graded by the Common terminology criteria for adverse event v4.0. (CTCAE v4.0). | from the beginning of radiotherapy up to 1 year after the 1st session.
  Current score for radiation pneumonitis according to symptoms and radiographic changes. Grade 0: No changes, Grade 1: Asymptomatic or mild respiratory symptoms, Grade 2: Moderate respiratory symptoms of pneumonitis (a severe cough) and radiographic changes (radiographic patches), Grade 3: Severe respiratory symptoms of pneumonitis, dense radiographic changes. Grade 4: Symptoms of acute respiratory failure requiring assisted ventilation or continuous oxygen. Grade 5: Death directly related to late effects of radiotherapy.
Pneumonitis graded by the Radiation Therapy Oncology Group score (RTOG) | from the beginning of radiotherapy up to 1 year after the 1st session.
  Current score for radiation pneumonitis according to symptoms and radiographic changes. Grade 0: No changes, Grade 1: Asymptomatic, only radiological or tomographic findings, Grade 2: Symptomatic, does not interfere with daily activities, Grade 3: Symptomatic, interferes with daily activities, requires supplemental oxygen. Grade 4: Threatens life, needing ventilator support. Grade 5: Severe pneumonitis with fatal outcome.

SECONDARY OUTCOMES:
Lung cancer-associated symptoms assessment | before the start of Radiotherapy, and at 6, 12, 24 and 48-weeks post-treatment.
  Symptoms are evaluated with the supplementary lung cancer-specific questionnaire of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (validated Mexican-Spanish version).
  It comprises 13 questions related to the assessment of dyspnoea, pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. The items scale ranges from 1 (Not at all) to 4 (Very much). The average of the items that contribute to the scale (raw score) is estimated and transformed so that scores range from 0 to 100. A higher scale score represents a higher level of symptoms.
Treatment-related side effects in lung cancer | before the start of Radiotherapy, and at 6, 12, 24 and 48-weeks post-treatment.
  Symptoms are evaluated with the supplementary lung cancer-specific questionnaire of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (validated Mexican-Spanish version).
  It comprises 13 questions related to the assessment of dyspnoea, pain, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. The items scale ranges from 1 (Not at all) to 4 (Very much). The average of the items that contribute to the scale (raw score) is estimated and transformed so that scores range from 0 to 100. A higher scale score represents a higher level of side-effects.
Cognitive functioning evaluated by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire | before the start of Radiotherapy, and at 6, 12, 24 and 48-weeks post-treatment.
  The cognitive functioning is evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires.
  It comprises two questions related to the assessment of short and long-term memory. The items scale ranges from 1 (Not at all) to 4 (Very much). The average of the items that contribute to the scale (raw score) is estimated and transformed so that scores range from 0 to 100. A higher scale score represents a healthy level of functioning.
Emotional Functioning evaluated by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire | before the start Radiotherapy, and at 6, 12, 24 and 48-weeks post-treatment
  The Emotional Functioning is evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires.
  It comprises four questions related to the assessment of depression, anxiety, irritability, and stress. The items scale ranges from 1 (Not at all) to 4 (Very much). The average of the items that contribute to the scale (raw score) is estimated and transformed so that the scores range from 0 to 100. A higher scale score represents a represents a healthy level of functioning.
Physical functioning evaluated by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire | before the start Radiotherapy, and at 6, 12, 24 and 48-weeks post-treatment.
  The Physical functioning is evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires.
  It comprises five questions related to self-sufficiency activities (eating, walking, laying in bed or completing simple chores). The items scale ranges from 1 (Not at all) to 4 (Very much). The average of the items that contribute to the scale (raw score) is estimated and transformed so that the scores range from 0 to 100. A higher scale score represents a represents a healthy level of functioning.
Role Functioning evaluated by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire | before the start Radiotherapy, and at 6, 12, 24 and 48-weeks post-treatment.
  The Role functioning is evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires.
  It comprises two questions related to daily activities (work and hobbies limitation). The items scale ranges from 1 (Not at all) to 4 (Very much). The average of the items that contribute to the scale (raw score) is estimated and transformed so that the scores range from 0 to 100. A higher scale score represents a represents a healthy level of functioning.
Social Functioning evaluated by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire | before the start Radiotherapy, and at 6, 12, 24 and 48-weeks post-treatment.
  The Social Functioning is evaluated using the validated Mexican-Spanish version of the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaires.
  It comprises two questions related to family life and social activities. The items scale ranges from 1 (Not at all) to 4 (Very much). The average of the items that contribute to the scale (raw score) is estimated and transformed so that the scores range from 0 to 100. A higher scale score represents a represents a healthy level of functioning.
Respiratory symptoms evaluation using St. George respiratory questionnaire | before the start Radiotherapy, and at 6, 12, 24 and 48-weeks post-treatment.
  Respiratory symptoms are evaluated using the St. George respiratory questionnaire validated to Mexican-Spanish version. It is a disease-specific instrument designed to measure the impact on overall health, daily life, and perceived well-being in patients with airways disease. Scores range from 0 to 100, with higher scores indicating more limitations.
Dyspnea assessment by the Borg Scale Dyspnea Index (BSDI) | before the start Radiotherapy, and at 6, 12, 24 and 48-weeks post-treatment.
  A system used to document the severity of the patient's shortness of breath using numbers anchored with verbal descriptions. This scale asks the patient to rate the dyspnea. It starts at number 0 where the breathing is causing no difficulty at all and progresses through to number 10 where the breathing difficulty is maximal.
Pulmonary function evaluation using spirometry test | before the start of Radiotherapy, and at 6, 12, 24 and 48-weeks post-treatment
  Spirometry measures the inhaled and exhaled air volume as a function of time using a forced expiratory maneuver.
Pulmonary function evaluation using diffusion lung capacity of carbon monoxide measurement (DLCO). | before the start of Radiotherapy and at 6, 12, 24 and 48-weeks post-treatment.
  Diffusion lung capacity of carbon monoxide (DLCO) test measures the conductance of gas transfer from inspired gas to the red blood cells.
Airway inflammatory response evaluation using the fraction of exhaled nitric oxide measurement (FeNO) | before the start of Radiotherapy, and at 6, 12, 24 and 48-weeks post-treatment.
  Nitric oxide concentration detected in the exhaled gas by chemiluminescence reported as particles per million.
Pulmonary function evaluation using Impulse oscillometry test (IOS) | before the start of Radiotherapy, and at 6, 12, 24 and 48-weeks post-treatment.
  Impulse oscillometry provides a rapid, noninvasive measure of airway impedance during normal tidal breathing.

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, MD MSc, Principal Investigator — Instituto Nacional de Cancerologia, Mexico
Locations (2):
- Mexico (2):
  - Instituto Nacional de Cancerologia, Mexico City
  - Instituto Nacional de Enfermedades Respiratorias, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
The data of the participants will be reported in the publication results.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: october 2021
Access Criteria: the information will be available after being published in an indexed journal, any information or data related to this study must be requested via e-mail with the researchers.

REFERENCES:
- [Result] Arrieta O, Guzman-de Alba E, Alba-Lopez LF, Acosta-Espinoza A, Alatorre-Alexander J, Alexander-Meza JF, Allende-Perez SR, Alvarado-Aguilar S, Araujo-Navarrete ME, Argote-Greene LM, Aquino-Mendoza CA, Astorga-Ramos AM, Austudillo-de la Vega H, Aviles-Salas A, Barajas-Figueroa LJ, Barroso-Quiroga N, Blake-Cerda M, Cabrera-Galeana PA, Calderillo-Ruiz G, Campos-Parra AD, Cano-Valdez AM, Capdeville-Garcia D, Castillo-Ortega G, Casillas-Suarez C, Castillo-Gonzalez P, Corona-Cruz JF, Correa-Acevedo ME, Cortez-Ramirez SS, de la Cruz-Vargas JA, de la Garza-Salazar JG, de la Mata-Moya MD, Dominguez-Flores ME, Dominguez-Malagon HR, Dominguez-Parra LM, Dominguez-Peregrina A, Duran-Alcocer J, Enriquez-Aceves MI, Elizondo-Rios A, Escobedo-Sanchez MD, de Villafranca PE, Flores-Cantisani A, Flores-Gutierrez JP, Franco-Marina F, Franco-Gonzalez EE, Franco-Topete RA, Fuentes-de la Pena H, Galicia-Amor S, Gallardo-Rincon D, Gamboa-Dominguez A, Garcia-Andreu J, Garcia-Cuellar CM, Garcia-Sancho-Figueroa MC, Garcia-Torrentera R, Gerson-Cwilich R, Gomez-Gonzalez A, Green-Schneeweiss L, Guillen-Nunez Mdel R, Gutierrez-Velazquez H, Ibarra-Perez C, Jimenez-Fuentes E, Juarez-Sanchez P, Juarez-Ramiro A, Kelly-Garcia J, Kuri-Exsome R, Lazaro-Leon JM, Leon-Rodriguez E, Llanos-Osuna S, Llanos-Osuna S, Loyola-Garcia U, Lopez-Gonzalez JS, Lopez y de Antunano FJ, Loustaunau-Andrade MA, Macedo-Perez EO, Machado-Villarroel L, Magallanes-Maciel M, Martinez-Barrera L, Martinez-Cedillo J, Martinez-Martinez G, Medina-Esparza A, Meneses-Garcia A, Mohar-Betancourt A, Morales Blanhir J, Morales-Gomez J, Motola-Kuba D, Najera-Cruz MP, Nunez-Valencia Cdel C, Ocampo-Ocampo MA, Ochoa-Vazquez MD, Olivares-Torres CA, Palomar-Lever A, Patino-Zarco M, Perez-Padilla R, Pena-Alonso YR, Perez-Romo AR, Aquilino Perez M, Pinaya-Ruiz PM, Pointevin-Chacon MA, Poot-Braga JJ, Posadas-Valay R, Ramirez-Marquez M, Reyes-Martinez I, Robledo-Pascual J, Rodriguez-Cid J, Rojas-Marin CE, Romero-Bielma E, Rubio-Gutierrez JE, Saenz-Frias JA, Salazar-Lezama MA, Sanchez-Lara K, Sansores Martinez R, Santillan-Doherty P, Alejandro-Silva J, Tellez-Becerra JL, Toledo-Buenrostro V, Torre-Bouscoulet L, Torecillas-Torres L, Torres M, Tovar-Guzman V, Turcott-Chaparro JG, Vazquez-Cortes JJ, Vazquez-Manriquez ME, Vilches-Cisneros N, Villegas-Elizondo JF, Zamboni MM, Zamora-Moreno J, Zinser-Sierra JW. [National consensus of diagnosis and treatment of non-small cell lung cancer]. Rev Invest Clin. 2013 Mar;65 Suppl 1:S5-84. Spanish. PMID 24459776
- [Result] Timmerman R, McGarry R, Yiannoutsos C, Papiez L, Tudor K, DeLuca J, Ewing M, Abdulrahman R, DesRosiers C, Williams M, Fletcher J. Excessive toxicity when treating central tumors in a phase II study of stereotactic body radiation therapy for medically inoperable early-stage lung cancer. J Clin Oncol. 2006 Oct 20;24(30):4833-9. doi: 10.1200/JCO.2006.07.5937. PMID 17050868
- [Result] Henkenberens C, Janssen S, Lavae-Mokhtari M, Leni K, Meyer A, Christiansen H, Bremer M, Dickgreber N. Inhalative steroids as an individual treatment in symptomatic lung cancer patients with radiation pneumonitis grade II after radiotherapy - a single-centre experience. Radiat Oncol. 2016 Feb 2;11:12. doi: 10.1186/s13014-016-0580-3. PMID 26830686
- [Result] Kim S, Oh IJ, Park SY, Song JH, Seon HJ, Kim YH, Yoon SH, Yu JY, Lee BR, Kim KS, Kim YC. Corticosteroid therapy against treatment-related pulmonary toxicities in patients with lung cancer. J Thorac Dis. 2014 Sep;6(9):1209-17. doi: 10.3978/j.issn.2072-1439.2014.07.16. PMID 25276362
- [Result] Ding NH, Li JJ, Sun LQ. Molecular mechanisms and treatment of radiation-induced lung fibrosis. Curr Drug Targets. 2013 Oct;14(11):1347-56. doi: 10.2174/13894501113149990198. PMID 23909719
- [Result] Williams JP, Johnston CJ, Finkelstein JN. Treatment for radiation-induced pulmonary late effects: spoiled for choice or looking in the wrong direction? Curr Drug Targets. 2010 Nov;11(11):1386-94. doi: 10.2174/1389450111009011386. PMID 20583979
- [Result] Daley-Yates PT. Inhaled corticosteroids: potency, dose equivalence and therapeutic index. Br J Clin Pharmacol. 2015 Sep;80(3):372-80. doi: 10.1111/bcp.12637. Epub 2015 May 28. PMID 25808113
- [Result] Leach C, Colice GL, Luskin A. Particle size of inhaled corticosteroids: does it matter? J Allergy Clin Immunol. 2009 Dec;124(6 Suppl):S88-93. doi: 10.1016/j.jaci.2009.09.050. PMID 19962042
- [Result] Bledsoe TJ, Nath SK, Decker RH. Radiation Pneumonitis. Clin Chest Med. 2017 Jun;38(2):201-208. doi: 10.1016/j.ccm.2016.12.004. Epub 2017 Mar 1. PMID 28477633
- [Result] Simone CB 2nd. Thoracic Radiation Normal Tissue Injury. Semin Radiat Oncol. 2017 Oct;27(4):370-377. doi: 10.1016/j.semradonc.2017.04.009. PMID 28865520
- [Result] Vallard A, Rancoule C, Le Floch H, Guy JB, Espenel S, Le Pechoux C, Deutsch E, Magne N, Chargari C. [Medical prevention and treatment of radiation-induced pulmonary complications]. Cancer Radiother. 2017 Aug;21(5):411-423. doi: 10.1016/j.canrad.2017.03.004. Epub 2017 Jun 5. French. PMID 28596060